CLINICAL TRIAL: NCT01880528
Title: A Double-Blind Pilot Study to Measure the Effect of Lisinopril vs. Placebo on Pulmonary Distress in Patients Receiving External Beam Radiotherapy to the Lung
Brief Title: Lisinopril in Reducing Shortness of Breath Caused by Radiation Therapy in Patients With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC1221; NCI-2013-01139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-008062; P30CA015083 (NIH)
Record Dates: First submitted 2013-06-15; First posted 2013-06-19 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dyspnea; Non-small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Dyspnea; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lisinopril) (Experimental): Beginning within 7 days of beginning radiation therapy, patients receive lisinopril PO QD on days 1-7.
  Interventions: Drug: lisinopril
- Arm II (placebo) (Placebo Comparator): Beginning within 7 days of beginning radiation therapy, patients receive placebo PO QD on days 1-7.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lisinopril — Given PO
  Other Names: Prinivil; Zestril
  Arms: Arm I (lisinopril)
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This pilot clinical trial studies lisinopril in reducing shortness of breath caused by radiation therapy in patients with lung cancer. Lisinopril may decrease the side effects caused by radiation therapy in patients with lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the adverse event profile of lisinopril, during and after external beam radiation therapy (RT) to the lung.

SECONDARY OBJECTIVES:

I. To explore the level of patient-reported acute respiratory distress (dyspnea) during and after external beam RT.

II. To explore the level of patient-reported symptoms during and after external beam RT.

III. To explore the impact of lisinopril treatment on patient quality of life (QOL) during and after external beam RT.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Beginning within 7 days of beginning radiation therapy, patients receive lisinopril orally (PO) once daily (QD) on days 1-7.

ARM II: Beginning within 7 days of beginning radiation therapy, patients receive placebo PO QD on days 1-7.

In both arms, treatment repeats every 7 days for until 3 months after completion of radiation therapy in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of small cell and non-small cell carcinoma of the lung receiving thoracic radiotherapy > 45 Gy, with volume of lung receiving 20 Gy or more (V20Gy) >= 20%
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 9.0 g/dL
* Creatinine clearance >= 30 mL/min as calculated using actual body weight and Cockroft Gault formula
* Initial physical exam with systolic blood pressure (BP) of > 100 mmHg and diastolic BP of > 60 mmHg
* Potassium within institutional normal limits
* Sodium within institutional normal limits
* Negative pregnancy test done =< 14 days prior to registration, for women of childbearing potential only
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment (e.g., maintenance or adjuvant chemotherapy or hormonal therapy) for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* History of prior radiation therapy treatment to the lungs or thorax
* Existing contraindications to angiotensin-converting enzyme (ACE) inhibitors such as hypersensitivity to ACE inhibitors, bilateral renal artery stenosis, angioedema, or previously documented adverse drug reaction to ACE inhibitors
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Use of ACE inhibitors (including lisinopril) or ACE receptor blockers (ARB) of any kind =< 90 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05-31 (Actual); Primary Completion 2013-06-05 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Miller, M.D., Study Chair — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Lisinopril): Beginning within 7 days of beginning radiation therapy, patients receive lisinopril PO QD.
- Arm II (Placebo): Beginning within 7 days of beginning radiation therapy, patients receive placebo PO QD.
Period: Overall Study
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
Started | 12 | 11
Completed (Evaluable for primary endpoint) | 11 | 10
Not Completed | 1 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo) | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Median (Full Range); unit: years] | 62.0 [49.0 to 87.0] | 62.0 [54.0 to 83.0] | 62.0 [49.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade 3 or Higher Hypotension, Acute Kidney Injury, Allergic Reaction, or Anaphylaxis, as Measured Using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0
Description: Incidence of grade 3 or higher hypotension, acute kidney injury, allergic reaction, or anaphylaxis, as measured using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. Descriptive statistics of frequency (percentage) will be used to summarize adverse event (AE) incidence and severity in the lisinopril and placebo arms separately.
Time Frame: Up to 3 months post-radiation therapy
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 10
percentage of patients | 0 | 0

2. Secondary Outcome: Acute Respiratory Distress (Dyspnea), Measured Using of the Maximum Score, at Any Time, of the Shortness of Breath Question (Item #4) on the LCSS (Worst Dyspnea Score)
Description: Acute respiratory distress (dyspnea), measured using of the maximum score, at any time, of the shortness of breath question (Item #4 "How much shortness of breath do you have?") on the Lung Cancer Symptom Scale (LCSS) (Worst Dyspnea Score). The LCSS tool contains 6 major symptoms associated with lung malignancies and their effect on overall symptomatic distress, functional activities, and global quality of life (QOL). The item scale ranges from 0-10 (0 = None; 10 = As much as it could be) where the LCSS scoring algorithm is applied to convert to a 0-100 point scale where 100 is best quality of life (QOL), for comparability. Patient scores range from 0 to 100, where 100 was best QOL (i.e. less pulmonary distress).
Time Frame: Up to 3 months post-radiation therapy
Population: Patients who completed the LCSS Item #4 at any time during the study are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 10
score on a scale | 77.5 (23.8) | 42.0 (27.8)
Statistical Analysis 1: Comparison: Arm I (Lisinopril) vs Arm II (Placebo); Test type: Superiority; p = 0.006, Kruskal-Wallis

3. Secondary Outcome: Experience Shortness of Breath During Exercise as Measured Using Item #3 on the Symptom Experience Questionnaire (SEQ) at Week 4
Description: Experience shortness of breath during exercise as measured using Item #3 ("Over the past week, did you experience shortness of breath when you exercise or exert yourself?") on the Symptom Experience Questionnaire (SEQ) at Baseline. The item scale ranges from 0-10 (0 = Not at all; 10 = As bad as it can be) where the SEQ scoring algorithm is applied to convert to a 0-100 point scale where 100 is best quality of life (QOL), for comparability.
Time Frame: At Week 4
Population: Patients who completed Item #3 on the SEQ at week 4 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
Number analyzed (Participants) | 3 | 7
score on a scale | 100 (0) | 68.6 (27.9)
Statistical Analysis 1: Comparison: Arm I (Lisinopril) vs Arm II (Placebo); Test type: Superiority; p = 0.0337, Kruskal-Wallis

4. Secondary Outcome: Quality of Life (Dyspnea When Climbing Stairs) Assessed Using Item #5 of the European Organization for Research on the Treatment of Cancer Lung Cancer Module Survey (EORTC-QLQ-LC13) at Week 4
Description: Dyspnea when climbing as measured using item #5 ("Were you short of breath when you climbed stairs?") of the EORTC-QLQ-LC13 at Week 4. The item scale ranges from 1-4 (1 = Not at all; 4 = Very Much) where the EORTC-QLQ-LC13 scoring algorithm is applied to convert to a 0-100 point scale where 100 is best quality of life (QOL), for comparability.
Time Frame: At Week 4
Population: Patients who completed item #5 on the EORTC-QLQ-LC13 at week 4 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 9
score on a scale | 83.3 (17.8) | 51.9 (33.8)
Statistical Analysis 1: Comparison: Arm I (Lisinopril) vs Arm II (Placebo); Test type: Superiority; p = 0.0427, Kruskal-Wallis

5. Secondary Outcome: Total LCSS Score as Measure by the Lung Cancer Symptom Scale (LCSS) at Week 4
Description: Total LCSS score as measured using the Lung Cancer Symptom Scale (LCSS) at Week 4. The item scale ranges from 0-10 (0 = None; 10 = As much as it could be) where the LCSS scoring algorithm is applied to convert to a 0-100 point scale where 100 is best quality of life (QOL), for comparability.
Time Frame: At Week 4
Population: Patients who completed the LCSS at week 4 are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 9
score on a scale | 83.8 (11.2) | 66.5 (17.0)
Statistical Analysis 1: Comparison: Arm I (Lisinopril) vs Arm II (Placebo); Test type: Superiority; p = 0.0237, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Up to 3 months post-radiation therapy
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients assessed for AEs and completed AE form. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Arm I (Lisinopril) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/12 | 1/10
Other Adverse Events (participants affected / at risk) | 11/12 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lisinopril) (N=12) | Arm II (Placebo) (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (4) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lisinopril) (N=12) | Arm II (Placebo) (N=10)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Fatigue (General disorders) | 1 (5) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (26) | 9 (32)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 5 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes